CLINICAL TRIAL: NCT03840460
Title: A Prospective Translational Tissue Collection Study in Early and Advanced Pancreatic Ductal Adenocarcinoma (PDAC) and Pancreatic Neuroendocrine Tumours (PanNETs) to Enable Further Disease Characterisation and the Development of Potential Predictive and Prognostic Biomarkers
Brief Title: A Prospective Translational Tissue Collection Study in Early and Advanced Pancreatic Ductal Adenocarcinoma and Pancreatic Neuroendocrine Tumours to Enable Further Disease Characterisation and the Development of Potential Predictive and Prognostic Biomarkers
Acronym: PaC-MAn
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4753
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The collected blood and tissue will undergo molecular analyses, including but not limited to, miRNA analysis, DNA and RNA sequencing, nanostring, real-time PCR and immunohistochemistry. Molecular analysis data will be correlated with clinical outcome data and allow characterization of subtypes in pancreatic cancer, considering both pancreatic ductal adenocarcinoma and pancreatic neuroendocrine tumours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreatic Cancer: Patients who are investigated for and subsequently diagnosed with early/advanced pancreatic adenocarcinoma or a precursor lesion or a pancreatic neuroendocrine tumour.

SUMMARY:
There are several types of early pre-cancerous lesions found in the pancreas which have the potential to develop into pancreatic cancer. Although different patients' pancreatic cancers or pre-cancerous pancreatic lesions have many similarities we believe that subtle differences can affect how they behave and therefore influence individual patient outcomes. Many factors may account for the differences seen in pancreatic lesion behaviour, for example molecular and genetic differences (the DNA and RNA present which control how a cell grows and divides), differences in how the immune system responds to the lesion, differences in the environment immediately around the lesion in the pancreas, known as the tumour microenvironment and differences in the micro-organisms which colonize a particular patient, known as their microbiota .

This project studies the molecular makeup of pancreatic lesions and their microenvironment at various stages (from pre-cancerous lesions all the way through to more advanced disease) to see if we can use this information to divide patients into different groups whose lesions may behave in similar ways. We will be trying to find out if there are molecular reasons why some patients respond to particular treatments when others do not, why some patients experience more toxicity with particular treatments and why some patients' disease behaves particularly aggressively when other patients' disease does not. We will also be investigating the particular micro-organisms colonizing individual patients to see if these impact a patient's outcome. Understanding what makes one person's pancreatic lesion behave differently to another's could lead to better treatment, where a personalized therapeutic strategy could be applied for every single patient.

DETAILED DESCRIPTION:
The main objective is to describe the incidence and distribution of tumour biomarkers, and to identify molecular subgroups from a multicentre series of patients who are investigated for and subsequently diagnosed with a pancreatic adenocarcinoma (PDAC) or a precursor lesion or a pancreatic neuroendocrine tumour.

The secondary objective is to determine disease control rate (CR, PR and SD >24 weeks), duration of response, progression free survival (PFS) and overall survival (OS) in locally advanced / metastatic patients or relapse free survival (RFS) and overall survival (OS) in early stage curative / pre-cursor lesion patients, associated with the identified molecular subtypes of PDAC pancreatic cancer and relevant anti-cancer therapies.

To identify molecular predictors of response or toxicity to standard of care anti-cancer therapies in PDAC/PanNET. The study also has a number of exploratory objectives listed below:

Depending on the number of patients assessable for each biomarker of interest and the prevalence of biomarker expression in the study population, exploratory endpoints of this study include:

1. Evaluation of the predictive value of biomarker expression (i.e. the ability of a biomarker to predict responsiveness or resistance to a specific anti-cancer treatment).
2. Evaluation of the prognostic value of biomarker expression (i.e. the ability of a biomarker to predict outcome regardless of a specific anti-cancer treatment).
3. Comparison of biomarker expression among IPMN, MCN, and pancreatic adenocarcinoma and evaluation of their prognostic value.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is being investigated or treated for pancreatic cancer or precursor lesions at The Royal Marsden Hospital and referring centres during the study period.
2. Patient has a histologically/cytologically confirmed diagnosis of pancreatic ductal adenocarcinoma, or pancreatic neuroendocrine tumour OR Patient has a tissue lesion suspicious for pancreatic cancer amenable to core needle biopsy or surgery and is clinically fit enough to undergo a tumour biopsy or surgery according to investigator assessment and local guidelines.
3. Patient is ≥ 18 years of age.
4. Patient can understand the patient information sheet and is able to provide written informed consent.
5. Patient has sufficient tissue and/or blood and/or urine and/or stool and/or saliva sampling for analysis as per the protocol.

Exclusion Criteria:

1. Patients who are not treated at all at The Royal Marsden Hospital or referring centre.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient is ≥ 18 years of age.
Study Population: early/advanced pancreatic adenocarcinoma or a precursor lesion or a pancreatic neuroendocrine tumour.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-01-10 (Estimated); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
to describe the incidence and distribution of biomarkers and identify molecular subtypes in a large, multi-centre, series of patients with pancreatic cancer and precursor lesions. | 4 years
  Blood, urine, stool, saliva, bile and tissue samples from patients undergoing a tissue biopsy or surgery for suspected or known pancreatic cancer will be collected

SECONDARY OUTCOMES:
To describe the incidence and distribution of biomarkers and identify molecular subtypes in a large, multi-centre, population of patients with pancreatic cancer or precursor lesions. | 4 years
  Molecular analyses including, but not limited to, miRNA analysis, DNA and RNA sequencing, nanostring, RT-PCR and immunohistochemistry will be carried out.
To identify molecular predictors of response or toxicity to standard of care anti-cancer therapies in PDAC/PanNET. | 4 years
  Blood, urine, stool, saliva, bile and tissue samples from patients undergoing a tissue biopsy or surgery for suspected or known pancreatic cancer will be collected. Molecular analyses including, but not limited to, miRNA analysis, DNA and RNA sequencing, nanostring, RT-PCR and immunohistochemistry will be carried out.

OTHER OUTCOMES:
Depending on the number of patients assessable for each biomarker of interest and the prevalence of biomarker expression in the study population, exploratory endpoints of this study include | 4 years
  evaluation of the predictive value of biomarker expression (i.e. the ability of a biomarker to predict responsiveness or resistance to a specific anti-cancer treatment).
Depending on the number of patients assessable for each biomarker of interest and the prevalence of biomarker expression in the study population, exploratory endpoints of this study include | 4 years
  evaluation of the prognostic value of biomarker expression (i.e. the ability of a biomarker to predict outcome regardless of a specific anti-cancer treatment).
Depending on the number of patients assessable for each biomarker of interest and the prevalence of biomarker expression in the study population, exploratory endpoints of this study include | 4 years
  comparison of biomarker expression among IPMN, MCN, and pancreatic adenocarcinoma and evaluation of their prognostic value.

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Study Chair — The Royal Marsden Hospital NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom